CLINICAL TRIAL: NCT03734029
Title: A Phase 3, Multicenter, Randomized, Open-label, Active Controlled Trial of DS-8201a, an Anti-HER2-antibody Drug Conjugate (ADC), Versus Treatment of Physician's Choice for HER2-low, Unresectable and/or Metastatic Breast Cancer Subjects
Brief Title: Trastuzumab Deruxtecan (DS-8201a) Versus Investigator's Choice for HER2-low Breast Cancer That Has Spread or Cannot be Surgically Removed [DESTINY-Breast04]
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U303; 2018-003069-33 (EudraCT Number); 184223 (Registry Identifier: JAPIC CTI); DESTINY-B04 (Other: Daiichi Sankyo and AstraZeneca)
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Anti-HER2-Antibody Drug Conjugate (ADC); Unresectable or Metastatic; Human epidermal growth factor receptor 2 (HER2)-low; DESTINY - Breast 04
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — trastuzumab deruxtecan; Capecitabine; eribulin; Gemcitabine; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Parallel model, randomized at a 2:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trastuzumab deruxtecan (Experimental): HER2-low, unresectable, and/or metastatic breast cancer participants previously treated with chemotherapy randomized to DS8201a
  Interventions: Drug: Trastuzumab deruxtecan (DS-8201a)
- Physician's Choice (Active Comparator): HER2-low, unresectable, and/or metastatic breast cancer participants previously treated with chemotherapy randomized to Physician's choice from the following options:
  * Capecitabine
  * Eribulin
  * Gemcitabine
  * Paclitaxel
  * Nab-paclitaxel
  Interventions: Drug: Capecitabine; Drug: Eribulin; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Trastuzumab deruxtecan (DS-8201a) — DS-8201a is a lyophilized powder reconstituted into a sterile aqueous solution (100 mg/5 mL) to be administered intravenously
  Other Names: DS-8201a
  Arms: Trastuzumab deruxtecan
Drug: Capecitabine — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Arms: Physician's Choice
Drug: Eribulin — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Arms: Physician's Choice
Drug: Gemcitabine — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Arms: Physician's Choice
Drug: Paclitaxel — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Arms: Physician's Choice
Drug: Nab-paclitaxel — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Arms: Physician's Choice

SUMMARY:
This study will compare DS-8201a to physician choice standard treatment.

Participants must have HER2-low breast cancer that has been treated before.

Participants' cancer:

* Cannot be removed by an operation
* Has spread to other parts of the body

DETAILED DESCRIPTION:
This is a randomized, 2-arm, Phase 3, open-label, multicenter study to compare the safety and efficacy of trastuzumab deruxtecan versus the physician's choice (2:1) in HER2-low, unresectable and/or metastatic breast cancer participants.

The Sponsor proposes to define a new HER2-low population in this trial including tumors with IHC 1+ and IHC 2+/ISH- HER2 expression.

ELIGIBILITY:
Inclusion Criteria:

* Is the age of majority in their country
* Has pathologically documented breast cancer that:

  1. Is unresectable or metastatic
  2. Has low-HER2 expression defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested)
  3. Is HR-positive or HR-negative
  4. Has progressed on, and would no longer benefit from, endocrine therapy
  5. Has been treated with 1 to 2 prior lines of chemotherapy/adjuvant in the recurrent or metastatic setting
  6. Was never previously HER2-positive (ICH 3+ or ISH+) on prior pathology testing (per American Society of Clinical Oncology-College of American Pathologists [ASCO-CAP] guidelines)
* Has documented radiologic progression (during or after most recent treatment)
* Has adequate archival tumor samples available or is wiling to provide fresh biopsies prior to randomization for:

  1. assessment of HER2 status
  2. assessment of post-treatment status
* Has at least 1 measurable lesion per Response Evaluation Criteria In Solid Tumors 1.1
* Has protocol-defined adequate cardiac, bone marrow, renal, hepatic and blood clotting functions
* Male and female participants of reproductive/childbearing potential, agrees to follow instructions for method(s) of contraception and agrees to avoid preserving ova or sperm for at least 4.5 months after treatment (or longer, per locally approved labels)

Exclusion Criteria:

* Is ineligible for all options in the physician's choice arm
* Has breast cancer ever assessed with high-HER2 expression
* Has previously been treated with any anti-HER2 therapy, including an antibody drug conjugate
* Has uncontrolled or significant cardiovascular disease
* Has spinal cord compression or clinically active central nervous system metastases
* Has history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
* Has any medical history or condition that per protocol or in the opinion of the investigator is inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2026-08-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (208):
- United States (38):
  - Ironwood Cancer & Research Centers - Chandler II, Chandler, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cancer Treatment Centers of America at Western Regional Medical Center, Goodyear, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Cancer Care Associates Medical Group, Inc. TORI, Redondo Beach, California
  - University of California at San Francisco (PARENT), San Francisco, California
  - Eastern Connecticut Hematology/Oncology Assoc., Norwich, Connecticut
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Sylvester Comprehensive Cancer Center - Deerfield Beach, Boca Raton, Florida
  - Florida Cancer Specialists (South Region), Fort Myers, Florida
  - Memorial Healthcare System MRH Cancer Center, Hollywood, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Moffitt Cancer Center -Tampa, Tampa, Florida
  - Cancer Treatment Centers of America-Georgia, Newnan, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Cancer Treatment Centers of America, Zion, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Touro Infirmary, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - New York University Medical Center, New York, New York
  - Memorial Sloan Kettering Hospital, New York, New York
  - Weill Cornell Medicine Breast Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - St Francis Hospital, Greenville, South Carolina
  - Brig Center for Cancer Care and Survivorship, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Tennessee Oncology - Skyline Satellite, Nashville, Tennessee
  - BloomTrials Clinical Research, LLC, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - University of Texas M. D. Anderson Cancer Center - Investigational Cancer Therapeutics, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Austria (5):
  - Medizinische Universität Innsbruck, Innsbruck
  - Kepler Universitätsklinikum, Linz
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - AKH - Medizinische Universität Wien (4305), Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - Grand Hôpital de Charleroi, Loverval
  - CHU UCL Namur, Namur
  - Centre Hospitalier Wallonie picarde - Site IMC, Tournai
- Canada (3):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology Clinical Research Program, Montreal, Quebec
- China (18):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Area Command of Chinese PLA, Fuzhou, Fujian
  - Sun Yat-sen Memorial hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia Hui
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (19):
  - Institut Paoli Calmettes, Marseille, Bouches-du-Rhône
  - Centre François Baclesse, Caen, Calvados
  - CARIO - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, Plérin, Cotes d'Armor
  - CHU Brest - Hôpital Morvan, Brest, Finistere
  - Institut Bergonié, Bordeaux, Gironde
  - Clinique Clementville, Montpellier, Herault
  - Institut Régional du Cancer de Montpellier, Montpellier, Herault
  - CRLCC Eugene Marquis, Rennes, Ille Et Vilaine
  - ICO - Site René Gauducheau, Saint-Herblain, Loire Atlantique
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay, Loiret
  - ICO - Site Paul Papin, Angers, Maine Et Loire
  - Centre Hospitalier Valenciennes, Valenciennes, Nord
  - Hôpital Saint-Louis - Paris, Paris, Paris
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Sarthe
  - Institut Sainte Catherine, Avignon, Vaculuse
  - Hôpital d'Instruction des Armees Begin*, Saint-Mandé, Val De Marne
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - Institut Curie - site de Paris, Paris
  - Hopital Tenon, Paris
- Germany (2):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum der Universitaet Muenchen - Campus Grosshardern, Munich, Bavaria
- Greece (9):
  - General Hospital of Athens "Alexandra", Athens
  - General Oncology Hospital of Kifissia " Agioi Anargyroi", Athens
  - Athens Medical Center, Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa
  - Bioclinic Thessaloniki, Thessaloniki
  - Euromedica General Clinic Thessaloniki, Thessaloniki
  - General Hospital Papageorgiou, Thessaloniki
  - Interbalkan Hospital of Thessaloniki, Thessaloniki
- Hungary (6):
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem, Debrecen
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Israel (8):
  - Rambam Health Care Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Azienda Ospedaliera Card. G. Panico, Tricase, Lecce
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliera Univ. Policlinico Gaspare Rodolico, Catania
  - Azienda Ospedaliero Universitaria Mater Domini-Campus Universitario, Catanzaro
  - IEO Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Ospedale degli Infermi, Rimini
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Japan (18):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - NHO Kyushu Cancer Center, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - NHO Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, Hyōgo
  - Hakuaikai Sagara Hospital, Kagoshima, Kagoshima-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - NHO Osaka National Hospital, Osaka, Osaka
  - Kindai University Hospital, Onohigashi, Osakasayama-shi
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Cancer Institute Hospital of JFCR, Kōtoku, Tokyo-To
  - Toranomon Hospital, Minatoku, Tokyo-To
  - Showa University Hospital, Shinagawa-Ku, Tokyo-To
- Portugal (10):
  - Hospital de Braga, Braga
  - Centro Hospitalar do Alto do Ave, EPE, Guimarães
  - Fundação Champalimaud, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saúde de Matosinhos, EPE (Hospital Pedro Hispano), Matosinhos Municipality
  - Centro Hospitalar do Porto, E.P.E. - Hospital de Santo António, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E - Hospital de São Sebastião, Santa Maria da Feira
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E, Vila Nova de Gaia
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, EPE, Vila Real
- Russia (3):
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - SBIH of Moscow City "Moscow City Oncology Hospital №62" of Moscow Healthcare Departement, Moscow
  - SBIH of Yaroslavl Region "Regional Clinical Oncological Hospital", Yaroslavl
- South Korea (11):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Inha University Hospital, Incheon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (18):
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Donostia, San Sebastián, Guipuzcoa
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital del Mar, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - MD Anderson Cancer Centre, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano de Oncologia IVO, Valencia
  - Hospital General Universitario de Valencia, Valencia
- Sweden (3):
  - Karolinska universitetssjukhuset - Solna, Solna
  - Länssjukhuset Sundsvall-Härnösand, Sundsvall
  - Akademiska Sjukhuset, Uppsala
- Switzerland (7):
  - Hirslanden Medical Center, Aarau
  - Universitaetsspital Basel, Basel
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Universitaetsspital Zuerich, Zurich
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (7):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Queen Mary University of London, London, Greater London
  - University College London Hospitals, London, Greater London
  - Royal Free Hospital, London, Greater London
  - Western General Hospital, Edinburgh, Lothian Region
  - Nottingham University Hospitals City Campus, Nottingham, Nottinghamshire
  - Royal Surrey County Hospital, Guildford, Surrey

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Result] Modi S, Jacot W, Yamashita T, Sohn J, Vidal M, Tokunaga E, Tsurutani J, Ueno NT, Prat A, Chae YS, Lee KS, Niikura N, Park YH, Xu B, Wang X, Gil-Gil M, Li W, Pierga JY, Im SA, Moore HCF, Rugo HS, Yerushalmi R, Zagouri F, Gombos A, Kim SB, Liu Q, Luo T, Saura C, Schmid P, Sun T, Gambhire D, Yung L, Wang Y, Singh J, Vitazka P, Meinhardt G, Harbeck N, Cameron DA; DESTINY-Breast04 Trial Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Low Advanced Breast Cancer. N Engl J Med. 2022 Jul 7;387(1):9-20. doi: 10.1056/NEJMoa2203690. Epub 2022 Jun 5. PMID 35665782
- [Derived] Modi S, Jacot W, Iwata H, Park YH, Vidal Losada M, Li W, Tsurutani J, Ueno NT, Zaman K, Prat A, Papazisis K, Rugo HS, Yamashita T, Harbeck N, Im SA, De Laurentiis M, Pierga JY, Wang X, Gombos A, Tokunaga E, Orbegoso Aguilar C, Yung L, Xiao F, Cheng Y, Cameron D. Trastuzumab deruxtecan in HER2-low metastatic breast cancer: long-term survival analysis of the randomized, phase 3 DESTINY-Breast04 trial. Nat Med. 2025 Dec;31(12):4205-4213. doi: 10.1038/s41591-025-03981-4. Epub 2025 Oct 8. PMID 41062831
- [Derived] Ueno NT, Cottone F, Dunton K, Jacot W, Yamashita T, Sohn J, Tokunaga E, Prat A, Tsurutani J, Park YH, Rugo HS, Xu B, Cardoso F, Mitri Z, Mahtani R, Aguilar CO, Xiao F, Harbeck N, Cameron DA, Modi S. Patient-reported outcomes from DESTINY-Breast04: trastuzumab deruxtecan versus physician's choice of chemotherapy in patients with HER2-low mBC. Oncologist. 2025 May 8;30(5):oyaf048. doi: 10.1093/oncolo/oyaf048. PMID 40349139
- [Derived] Yamashita T, Sohn JH, Tokunaga E, Niikura N, Park YH, Lee KS, Chae YS, Xu B, Wang X, Im SA, Li W, Lu YS, Aguilar CO, Nishijima S, Nishiyama Y, Sugihara M, Modi S, Tsurutani J. Trastuzumab deruxtecan versus treatment of physician's choice in previously treated Asian patients with HER2-low unresectable/metastatic breast cancer: subgroup analysis of the DESTINY-Breast04 study. Breast Cancer. 2024 Sep;31(5):858-868. doi: 10.1007/s12282-024-01600-7. Epub 2024 Jun 17. PMID 38884900
- [Derived] Ma R, Shi Y, Yan R, Yin S, Bu H, Huang J. Efficacy and safety of trastuzumab deruxtecan in treating human epidermal growth factor receptor 2-low/positive advanced breast cancer:A meta-analysis of randomized controlled trials. Crit Rev Oncol Hematol. 2024 Apr;196:104305. doi: 10.1016/j.critrevonc.2024.104305. Epub 2024 Mar 3. PMID 38442809
- [Derived] Jhaveri K, Eli LD, Wildiers H, Hurvitz SA, Guerrero-Zotano A, Unni N, Brufsky A, Park H, Waisman J, Yang ES, Spanggaard I, Reid S, Burkard ME, Vinayak S, Prat A, Arnedos M, Bidard FC, Loi S, Crown J, Bhave M, Piha-Paul SA, Suga JM, Chia S, Saura C, Garcia-Saenz JA, Gambardella V, de Miguel MJ, Gal-Yam EN, Rapael A, Stemmer SM, Ma C, Hanker AB, Ye D, Goldman JW, Bose R, Peterson L, Bell JSK, Frazier A, DiPrimeo D, Wong A, Arteaga CL, Solit DB. Neratinib + fulvestrant + trastuzumab for HR-positive, HER2-negative, HER2-mutant metastatic breast cancer: outcomes and biomarker analysis from the SUMMIT trial. Ann Oncol. 2023 Oct;34(10):885-898. doi: 10.1016/j.annonc.2023.08.003. Epub 2023 Aug 18. PMID 37597578
- [Derived] Rugo HS, Crossno CL, Gesthalter YB, Kelley K, Moore HB, Rimawi MF, Westbrook KE, Buys SS. Real-World Perspectives and Practices for Pneumonitis/Interstitial Lung Disease Associated With Trastuzumab Deruxtecan Use in Human Epidermal Growth Factor Receptor 2-Expressing Metastatic Breast Cancer. JCO Oncol Pract. 2023 Aug;19(8):539-546. doi: 10.1200/OP.22.00480. Epub 2023 May 19. PMID 37207306
- [Derived] Narayan P, Dilawari A, Osgood C, Feng Z, Bloomquist E, Pierce WF, Jafri S, Kalavar S, Kondratovich M, Jha P, Ghosh S, Tang S, Pazdur R, Beaver JA, Amiri-Kordestani L. US Food and Drug Administration Approval Summary: Fam-Trastuzumab Deruxtecan-nxki for Human Epidermal Growth Factor Receptor 2-Low Unresectable or Metastatic Breast Cancer. J Clin Oncol. 2023 Apr 10;41(11):2108-2116. doi: 10.1200/JCO.22.02447. Epub 2023 Feb 13. PMID 36780610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 557 participants were enrolled and randomized to treatment at 161 study sites in the United States (27 study sites), Japan (18 sites), France (16 sites), China (15 sites), Italy (13 sites), Spain (12 sites), Greece (8 sites), Portugal (8 sites), Republic of Korea (8 sites), Israel (6 sites), Switzerland (6 sites), Austria (4 sites), Belgium (4 sites), Russia (3 sites), Sweden (3 sites), Taiwan (3 sites), Unted Kingdom (3 sites), Canada (2 sites), and Hungary (2 sites).
Pre-assignment Details: All participants had been previously treated with at least 1 and no more than 2 prior lines of chemotherapy in the recurrent or metastatic setting. The treatment chosen for the Physician's Choice arm was based on the label approved in the country of drug administration. The Physician's Choice group was combined to ensure an appropriate sample size for the comparator group.
Groups:
- Trastuzumab Deruxtecan (T-DXd): Participants with HER2-low, unresectable, and/or metastatic breast cancer who were previously treated with chemotherapy were randomized to receive an intravenous infusion of DS8201a (initial dose of 5.4 mg/kg) over approximately 90 minutes. If there was no infusion-related reaction (IRR), T-DXd doses after the initial dose of 5.4 mg/kg were infused over a minimum of 30 minutes.
- Physician's Choice: Participants with HER2-low, unresectable, and/or metastatic breast cancer who were previously treated with chemotherapy and randomized to a physician's choice (capecitabine, eribulin, gemcitabine, paclitaxel, and nab-paclitaxel) in which the dose, regimen, administration, and dose modification followed the label approved in the country of drug administration or the National Comprehensive Cancer Network guidelines.
Period: Overall Study
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Started | 373 | 184
Full Analysis Set (All Randomized Patients) | 373 | 184
Safety Analysis Set (All Randomized Patients Who Received at Least 1 Dose of Study Treatment) | 371 | 172
Completed (Ongoing as of 11 Jan 2022) | 58 | 3
Not Completed | 315 | 181
Not completed — Progressive disease as per RECIST v1.1 | 220 | 130
Not completed — Adverse Event | 60 | 14
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Clinical progression by investigator | 10 | 8
Not completed — Death | 5 | 2
Not completed — Physician Decision | 4 | 3
Not completed — Other | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Randomized, but not treated | 2 | 12

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Full Analysis Set. The Full Analysis Set included all participants randomized into the study, including those who did not receive a dose of study treatment. Participants were analyzed according to the treatments and strata assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice | Total
Number analyzed (Participants) | 373 | 184 | 557
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 290 | 136 | 426
  >=65 years | 83 | 48 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.6) | 56.5 (11.5) | 56.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 371 | 184 | 555
  Male | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 176 | 91 | 267
  Black or African American | 7 | 3 | 10
  Asian | 151 | 72 | 223
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Other | 38 | 17 | 55
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Blinded Independent Central Review (BICR) in the Hormone Receptor-Positive Cohort in Participants With HER2-low Breast Cancer
Description: Progression-free survival (PFS), defined as at least a 20% increase in the sum of diameters of target lesions, was assessed from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever came first. PFS was based on blinded independent central review (BICR) in the hormone receptor-positive cohort according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.1. Median PFS was from Kaplan-Meier analysis. Confidence interval for median was computed using the Brookmeyer-Crowley method.
Time Frame: From the date of randomization to the earliest date of the first objective documentation of radiographic disease progression or death due to any cause, up to approximately 3 years
Population: Progression-free survival (PFS) was assessed in the Hormone Receptor-Positive cohort of Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 331 | 163
months | 10.1 [9.5 to 11.5] | 5.4 [4.4 to 7.1]
Statistical Analysis 1: Comparison: Trastuzumab Deruxtecan (T-DXd) vs Physician's Choice; Test type: Superiority; p < 0.0001, Log Rank — Two-sided p-value from stratified log-rank test, Hazard ratio and 95% CI from stratified Cox proportional hazards model using stratification factors: HER2 status, number of prior lines of chemotherapy, hormone Receptor/CDK status, as defined by IXRS; Cox Proportional Hazard = 0.5085, 95% CI 2-sided [0.4012 to 0.6444]

2. Secondary Outcome: Progression-free Survival (PFS) Based on Blinded Independent Central Review (BICR) in Participants With HER2-low Breast Cancer (All Patients) Regardless of Hormone Receptor Status
Description: Progression-free survival (PFS), defined as at least a 20% increase in the sum of diameters of target lesions, was assessed from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever came first. PFS was based on blinded independent central review (BICR) according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.1. Median PFS was from Kaplan-Meier analysis. Confidence interval for median was computed using the Brookmeyer-Crowley method.
Time Frame: as for outcome 1
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 373 | 184
months | 9.9 [9.0 to 11.3] | 5.1 [4.2 to 6.8]

3. Secondary Outcome: Progression-free Survival Based on Investigator Assessment in the Hormone Receptor-Positive Cohort in Participants With HER2-low Breast Cancer
Description: Progression-free survival (PFS), defined as at least a 20% increase in the sum of diameters of target lesions, was assessed from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever came first. PFS was based on investigator assessment in the hormone receptor-positive cohort according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.1. Median PFS was from Kaplan-Meier analysis. Confidence interval for median was computed using the Brookmeyer-Crowley method.
Time Frame: as for outcome 1
Population: Progression-free survival (PFS) was assessed in the Hormone Receptor-Positive cohort of Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 331 | 163
months | 9.6 [8.4 to 10.0] | 4.2 [3.4 to 4.9]

4. Secondary Outcome: Progression-free Survival Based on Investigator Assessment in Participants With HER2-low Breast Cancer (All Patients)
Description: Progression-free survival (PFS), defined as at least a 20% increase in the sum of diameters of target lesions, was assessed from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever came first. PFS was based on investigator assessment according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.1. Median PFS was from Kaplan-Meier analysis. Confidence interval for median was computed using the Brookmeyer-Crowley method.
Time Frame: as for outcome 1
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 373 | 184
months | 8.8 [8.3 to 9.8] | 4.2 [3.0 to 4.5]

5. Secondary Outcome: Overall Survival (OS) in the Hormone Receptor-Positive Cohort in Participants With HER2-low Breast Cancer
Description: Overall survival (OS) was defined as the time from the date of randomization to the date of death due to any cause. If there was no death reported for a participant before the data cutoff for OS analysis, OS was censored at the last contact date at which the participant was known to be alive.
Time Frame: From the date of randomization up to the date of death due to any cause, up to approximately 3 years
Population: Overall survival (OS) was assessed in the Hormone Receptor-Positive cohort of Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 331 | 163
months | 23.9 [20.8 to 24.8] | 17.5 [15.2 to 22.4]

6. Secondary Outcome: Number of Overall Survival Events (Deaths)
Time Frame: From the date of randomization up to the date of death due to any cause, up to approximately 3 years
Population: Overall survival events (deaths) were analyzed in the Full Analysis Set (defined as all randomized participants).
Measure: Number; unit: events (deaths)
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 373 | 184
events (deaths) | 149 | 90

7. Secondary Outcome: Overall Survival (OS) in All Patients
Description: as for outcome 5
Time Frame: From the date of randomization up to the date of death due to any cause, up to approximately 3 years
Population: Overall survival (OS) was assessed in the Full Analysis Set (defined as all randomized participants).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 373 | 184
months | 23.4 [20.0 to 24.8] | 16.8 [14.5 to 20.0]

8. Secondary Outcome: Best Overall Response and Confirmed Objective Response Rate (ORR) in the Hormone Receptor-Positive Cohort in Participants With HER2-low Breast Cancer
Description: Best overall response rate and confirmed objective response rate (ORR) were assessed by blinded independent central review (BICR) and investigator assessment. Complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions. Confirmed ORR was defined as the number of participants with complete and partial responses and confirmed by a second assessment.
Time Frame: From screening and every 6 weeks up to withdrawal of subject consent, progressive disease (PD), or unacceptable toxicity, up to approximately 3 years
Population: Best overall response and confirmed objective response rate were assessed in the Hormone Receptor-Positive cohort of Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 331 | 163
Participants
  BICR: Complete response | 12 | 1
  BICR: Partial response | 164 | 26
  BICR: Stable disease | 115 | 81
  BICR: Progressive disease | 26 | 34
  BICR: Not evaluable | 14 | 21
  Investigator: Complete response | 5 | 0
  Investigator: Partial response | 163 | 30
  Investigator: Stable disease | 124 | 80
  Investigator: Progressive disease | 28 | 34
  Investigator: Not evaluable | 11 | 19
  BICR: Confirmed Objective response rate | 175 | 27
  Investigator: Confirmed Objective response rate | 168 | 30

9. Secondary Outcome: Best Overall Response and Confirmed Objective Response Rate (ORR) in Participants With HER2-low Breast Cancer (All Patients)
Description: as for outcome 8
Time Frame: as for outcome 8
Population: Best overall response and confirmed objective response rate were assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 373 | 184
Participants
  BICR: Complete response | 13 | 2
  BICR: Partial response | 183 | 28
  BICR: Stable disease | 129 | 91
  BICR: Progressive disease | 31 | 41
  BICR: Not evaluable | 17 | 22
  Investigator: Complete response | 6 | 0
  Investigator: Partial response | 187 | 31
  Investigator: Stable disease | 135 | 93
  Investigator: Progressive disease | 32 | 40
  Investigator: Not evaluable | 13 | 20
  BICR: Confirmed Objective response rate | 195 | 30
  Investigator: Confirmed Objective response rate | 193 | 31

10. Secondary Outcome: Duration of Response in the Hormone Receptor-Positive Cohort in Participants With HER2-low Breast Cancer
Description: Duration of Response (DoR) is defined as the date of the first documented objective response (complete response [CR] or partial response [PR]) to the first documented disease progression or death, whichever occurs first. DoR was based on blinded independent central review (BICR) and investigator assessment. Median was from Kaplan-Meier estimate. Confidence interval for median was computed using the Brookmeyer-Crowley method.
Time Frame: From the date of the first documented objective response (CR or PR) to the first documented disease progression or death, whichever occurs first, up to approximately 3 years
Population: Duration of response was assessed in the Hormone Receptor-Positive cohort of Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 331 | 163
months
  BICR: DoR | 10.7 [8.5 to 13.7] | 6.8 [6.5 to 9.9]
  Investigator: DoR | 8.3 [7.1 to 11.1] | 5.6 [3.6 to 6.8]

11. Secondary Outcome: Duration of Response in Participants With HER2-low Breast Cancer (All Patients)
Description: as for outcome 10
Time Frame: as for outcome 10
Population: Duration of response was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 373 | 184
months
  BICR: DoR | 10.7 [8.5 to 13.2] | 6.8 [6.0 to 9.9]
  Investigator: DoR | 8.3 [7.0 to 9.9] | 5.6 [3.7 to 6.6]

12. Other Pre Specified Outcome: All-Cause Mortality
Description: All-cause mortality is defined as all anticipated and unanticipated deaths due to any cause, with the number and frequency of such events by arm or comparison group of the clinical study.
Time Frame: From the date of randomization up to the date of death due to any cause, up to approximately 3 years
Population: All-cause mortality was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
Number analyzed (Participants) | 371 | 172
Participants | 148 | 88

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of signing the main informed consent form up to 40 days (+7 days) after the last treatment, whether observed by the investigator or reported by the participant, up to approximately 3 years in the Safety Analysis Set.
Description: All-cause mortality was assessed in all participants who were randomized (Full Analysis Set). Please refer to the other prespecified outcome measure that also reports all-cause mortality from the Safety Analysis Set. Other AEs and SAEs were assessed in the Safety Analysis Set. The Physician's Choice (PC) treatment was based on the label approved in each country. As prespecified in the protocol for safety analysis, the PC group was combined for an appropriate sample size for the comparator group.
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Physician's Choice
All-Cause Mortality (participants affected / at risk) | 149/373 | 90/184
Serious Adverse Events (participants affected / at risk) | 103/371 | 43/172
Other Adverse Events (participants affected / at risk) | 366/371 | 167/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Deruxtecan (T-DXd) (N=371) | Physician's Choice (N=172)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 4
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 0
Disease progression (General disorders) | 2 | 2
Asthenia (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 1
Sepsis (Infections and infestations) | 5 | 0
COVID-19 (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Urosepsis (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 5
Medication error (Injury, poisoning and procedural complications) | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Social problem (Social circumstances) | 1 | 0
Embolism (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Superior vena cava occlusion (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Deruxtecan (T-DXd) (N=371) | Physician's Choice (N=172)
Anaemia (Blood and lymphatic system disorders) | 137 | 44
Neutropenia (Blood and lymphatic system disorders) | 49 | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 4
Nausea (Gastrointestinal disorders) | 281 | 52
Vomiting (Gastrointestinal disorders) | 148 | 23
Constipation (Gastrointestinal disorders) | 124 | 38
Diarrhoea (Gastrointestinal disorders) | 100 | 38
Stomatitis (Gastrointestinal disorders) | 41 | 17
Abdominal pain (Gastrointestinal disorders) | 35 | 8
Dyspepsia (Gastrointestinal disorders) | 34 | 11
Abdominal pain upper (Gastrointestinal disorders) | 31 | 13
Dry mouth (Gastrointestinal disorders) | 26 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 | 3
Abdominal distension (Gastrointestinal disorders) | 20 | 5
Fatigue (General disorders) | 110 | 49
Asthenia (General disorders) | 69 | 25
Pyrexia (General disorders) | 42 | 22
Malaise (General disorders) | 33 | 10
Oedema peripheral (General disorders) | 24 | 10
Urinary tract infection (Infections and infestations) | 27 | 6
Aspartate aminotransferase increased (Investigations) | 92 | 42
Neutrophil count decreased (Investigations) | 81 | 61
White blood cell count decreased (Investigations) | 78 | 49
Alanine aminotransferase increased (Investigations) | 75 | 43
Platelet count decreased (Investigations) | 72 | 12
Weight decreased (Investigations) | 59 | 14
Blood alkaline phosphatase increased (Investigations) | 36 | 5
Lymphocyte count decreased (Investigations) | 29 | 12
Blood bilirubin increased (Investigations) | 25 | 7
Gamma-glutamyltransferase increased (Investigations) | 20 | 8
Blood lactate dehydrogenase increased (Investigations) | 19 | 9
Decreased appetite (Metabolism and nutrition disorders) | 118 | 33
Hypokalaemia (Metabolism and nutrition disorders) | 38 | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 32 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 19 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 16
Headache (Nervous system disorders) | 53 | 11
Dysgeusia (Nervous system disorders) | 37 | 16
Dizziness (Nervous system disorders) | 32 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 18 | 19
Neuropathy peripheral (Nervous system disorders) | 13 | 16
Paraesthesia (Nervous system disorders) | 8 | 9
Insomnia (Psychiatric disorders) | 24 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 14
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 21 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 147 | 57
Rash (Skin and subcutaneous tissue disorders) | 24 | 9
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03734029/Prot_SAP_000.pdf